CLINICAL TRIAL: NCT01816581
Title: Prospective, Randomized Clinical Pilot Study: Oral Opiate Targin In Treatment Of Postoperative Pain After Major Cardiac Surgery
Brief Title: Oral Oxycodone After Major Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Kurt Rutzler, senior staff physician, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1043/2010
Record Dates: First submitted 2013-03-15; First posted 2013-03-22 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Heart; Dysfunction Postoperative, Cardiac Surgery
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Targin/OxyNorm (Active Comparator): Patients randomized to this study arm will receive Targin as basis pain medication and additional OxyNorm (Oxycodone), if requested by the patients.
  Interventions: Drug: Targin; Drug: Oxynorm
- PCA (Active Comparator): Patients randomized to this group will receive a PCA pump with morphine. The basic rate is 0.3 mg/h. Patients will be allowed to administer 1 mg each five minutes after a vesting period of five minutes, if subjectively needed.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Targin
  Other Names: Oxycodonhydrochlorid and naloxone hydrochloride dihydrate
  Arms: Targin/OxyNorm
Drug: Oxynorm
  Other Names: oral medication consisting of Oxycodonhydrochlorid
  Arms: Targin/OxyNorm
Drug: Morphine
  Arms: PCA

SUMMARY:
Postoperative pain and analgesic treatment still remains a challenge in daily perioperative medicine. Skin incisions, intraoperative tissue retraction and -dissection, intravasal cannulations and drainages, sternotomy and pericardiotomy are the most important reasons for postoperative pain. Poorly controlled pain can contribute directly or indirectly to postoperative complications, such as myocardial ischemia, pulmonary dysfunction like hypoventilation, pneumonia and atelectasis, a delayed return of gastrointestinal function and decreased mobility. In addition, prolonged acute pain also results in chronic pain.

Opioids are internationally recognized as the golden standard in the treatment of acute postoperative pain. On one side, the high potency of opioids in pain relief is clearly undisputed, but on the other hand, the administration of opioids is associated with nausea, vomiting, sedation and with the development of bowel dysfunction, which encompasses symptoms including bloating, abdominal spasm, cramps and constipation. Opioid-induced constipation is a frequently reported adverse effect and sometimes requires discontinuation of therapy, which results in analgesic under-treatment, severely impairing quality of life. However, there are many different regimes for the treatment of postoperative pain using opioids. Patient-controlled analgesia (PCA) using morphine is widely used, but requires trained staff and expensive equipment. Once patients are able to tolerate oral medications, the oral route is preferred postoperatively because it is more convenient, noninvasive and less expensive.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 90 years
* ASA physical status 1-3
* Elective major cardiac surgery requiring sternotomy
* Oral and written consent
* Postoperative extubation within four hours after arrival at the ICU
* Cognitive ability in the use of the PCA pump and the VAS

Exclusion Criteria:

* Chronic use of opioids in the last three months
* Chronic use of tranquilizer or pain medications
* Hypersensitivity against opioids
* Use of monoamine oxidase inhibitors in the last two weeks before surgery
* Alcohol or drug abuse
* Renal dysfunction (GFR < 30 or necessity of dialysis)
* Liver Dysfunction defined as Child-Pugh-Score 7-15
* Ejection fraction (EF< 40%)
* Malabsorption syndrome
* Neurologic or cognitive dysfunction
* Pregnancy
* Participation in another clinical trial
* Severe respiratory depression with hypoxia and/or hypercapnia
* Severe chronic obstructive pulmonary disease
* Severe bronchial asthma
* Non-opioid induced paralytic ileus
* Risk of seizures

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-07; Primary Completion 2012-05 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
total opioid dosage in terms of so-called morphine equivalents | 3 days
  total administrated opioid dosage during 3 days after surgery

SECONDARY OUTCOMES:
VAS pain score | 3 days
  Pain Scores on the Visual Analog Scale (0-100)
level of sedation | 3 days
  Level of Sedation using the Ramsey Sedation Score.
rate of spontaneous breathing | 3 days
  spontaneous breathing rate per minute
possible side effects | 3 days
  open documentation of any side effects like dizziness, vomiting, allergic reaction
in hospital stay | 1 month
ICU stay | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Ruetzler K, Blome CJ, Nabecker S, Makarova N, Fischer H, Rinoesl H, Goliasch G, Sessler DI, Koinig H. A randomised trial of oral versus intravenous opioids for treatment of pain after cardiac surgery. J Anesth. 2014 Aug;28(4):580-6. doi: 10.1007/s00540-013-1770-x. Epub 2013 Dec 28. PMID 24375220